CLINICAL TRIAL: NCT04342026
Title: Role of the Environment and Endocrine Disruptors in Child Cryptorchidism
Acronym: CRYPTENV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0544
Record Dates: First submitted 2020-03-20; First posted 2020-04-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cryptorchidism
Keywords: Cryptorchidism; environmental exposition; endocrine disruptors
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parent of patient with cryptorchidism: parent exposition of endocrine disruptors
  Interventions: Other: Measure of the exposure of parent of male with /without cryptorchidism to endocrine disruptors
- Parent of patient without cryptorchidism: Parent exposition of endocrine disruptors
  Interventions: Other: Measure of the exposure of parent of male with /without cryptorchidism to endocrine disruptors

INTERVENTIONS:
Other: Measure of the exposure of parent of male with /without cryptorchidism to endocrine disruptors — Measure of the exposure of parent of patient with/without cryptorchidism to endocrine disruptors (job exposure, during pregnancy)

SUMMARY:
Cryptorchidism is the most frequent congenital defect of the male newborn. It requires surgery in childhood, increases the risk of fertility disorders and cancer. As a major public health objective, it's the subject of numerous recommendations. Its frequency is increasing in some countries faster than a single genetic cause could not explain it. It may occurs in a geographic cluster. The cause of cryptorchidism involves genetic, hormonal and environmental factors. Animal studies suggest that endocrine disruptors interfere with fetal testicular migration. The aim of the study is to find out if some environmental exposition may be associated with cryptorchidism.

DETAILED DESCRIPTION:
Cryptorchidism is the most frequent congenital defect of the male newborn. It requires surgery in childhood, increases the risk of fertility disorders and cancer. As a major public health objective, it's the subject of numerous recommendations. Its frequency is increasing in some countries faster than a single genetic cause could not explain it. It may occurs in a geographic cluster. The cause of cryptorchidism involves genetic, hormonal and environmental factors. Animal studies suggest that endocrine disruptors interfere with fetal testicular migration. The aim of the study is to find out if some environmental exposition may be associated with cryptorchidism.

ELIGIBILITY:
Inclusion criteria:

- Parents of male children from the neonatal period to 18 years of age (during surgery) with cryptorchidism

Exclusion criteria:

* Parents of children without endocrine disease. (adrenal, hypothalamic-pituitary, phosphocalcic, thyroid, diabetes, etc.)
* Parents of children without an associated genital or urinary defect (hypospadias, micropenis, renal and bladder abnormalities)
* Testicular Ectopia (testis outside of normal migration path)
* Anorchidism and evanescent testicles, united or bilateral
* Abnormalities of the abdominal wall (laparoschisis, omphalocele, Prune Belly)
* Cryptorchidism integrating in the context of a polymalformative syndrome, including neurological.

Ages: 1 Month to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Parent of patient with cryptorchidism
Sampling Method: Probability Sample
Enrollment: 1452 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
frequency of the job exposure of the parents of endocrine disruptors | 1 day
  Measure of the frequency of endocrine disruptors assessed by european questionary QLK4-1999-01422 (simplified version )

SECONDARY OUTCOMES:
comparison of cryptorchid and non-cryptorchid children born to parents with isolated exposure vs multiple exposures | 1 day
  Assessement by the Job-exposure matrix EDC (Environment disrupting chemicals)
Comparison of frequencies of exposure to endocrine disruptors (Environmental Disrupting Chemicals) in parents giving birth to a congenital cryptorchid child vs child not cryptorchid at birth but with secondary cryptorchidism. | 1 day
  presence of cryptorchidism at birth or secondarily
identify food exposure criteria (phytoestrogen or EDC pesticides) associated with the presence of a cryptorchid. | 1 day
  parents will be asked about their diet
Constitution of collection of biological samples from children with non-palpable bilateral cryptorchidism | 1 day
  The aim is only to make a collection of blood samples. Anonymous samples will be used later in order to improve knowledge of the cryptorchidism.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France